CLINICAL TRIAL: NCT05512767
Title: Effects of a Pneumatic Compression Device in Post-Chemoradiation Head and Neck Cancer Population
Brief Title: A Pneumatic Compression Device for the Treatment of Lymphedema in Patients With Stage II-IV Head and Neck Cancer After Chemoradiation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI retired and study not moving forward
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-003342; NCI-2022-06767 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-08-17; First posted 2022-08-23 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Clinical Stage II HPV-Mediated (p16-pos) Oropharyngeal Carcinoma; Clinical Stage III HPV-Mediated (p16-pos) Oropharyngeal Carcinoma; Clinical Stage IV HPV-Mediated (p16-pos)Oropharyngeal Carcinoma; Head and Neck Carcinoma; Stage II Hypopharyngeal Carcinoma AJCC v8; Stage II Laryngeal Cancer AJCC v8; Stage II Lip and Oral Cavity Cancer AJCC v8; Stage II Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Practice Guidelines as Topic; Standard of Care; X-Rays; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group I (pneumatic therapy, lymphedema management) (Experimental): Patients undergo 32 minute treatments twice daily for 12 weeks using the FlexiTouch Plus System and treatment with a lymphedema therapist weekly on weeks 2-11. Patients undergo nasolaryngoscopy and videofluoroscopic swallow study at baseline.
  Interventions: Other: Consensus Auditory-Perceptual Evaluation of Voice; Procedure: Diagnostic Imaging; Other: Lymphedema Management; Procedure: Modified Barium Swallow; Procedure: Nasopharyngeal Laryngoscopy; Device: Pneumatic Compression Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Voice Handicap Index-10
- Group II (standard of care, lymphedema management) (Active Comparator): Patients undergo standard of care self-manual lymphatic drainage (technique instructions provided) twice daily for 12 weeks and treatment with a lymphedema therapist weekly on weeks 2-11. Patients undergo nasolaryngoscopy and videofluoroscopic swallow study at baseline.
  Interventions: Other: Best Practice; Other: Consensus Auditory-Perceptual Evaluation of Voice; Procedure: Diagnostic Imaging; Other: Lymphedema Management; Procedure: Modified Barium Swallow; Procedure: Nasopharyngeal Laryngoscopy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Voice Handicap Index-10

INTERVENTIONS:
Other: Best Practice — Undergo self-manual lymphatic drainage
  Other Names: standard of care; standard therapy
  Arms: Group II (standard of care, lymphedema management)
Other: Consensus Auditory-Perceptual Evaluation of Voice — Ancillary studies
  Other Names: CAPE-V; Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V)
Procedure: Diagnostic Imaging — Undergo photographs of face and neck
  Other Names: Medical Imaging
Other: Lymphedema Management — Undergo skilled lymphedema treatment by a therapist
Procedure: Modified Barium Swallow — Undergo swallow study
  Other Names: MBS; VFSS; Videofluoroscopic Swallowing Study
Procedure: Nasopharyngeal Laryngoscopy — Undergo Nasolaryngoscopy
Device: Pneumatic Compression Therapy — Undergo compression therapy - Flexitouch Plus System is an advanced pneumatic compression device (APCD) that consists of a 2-piece garment that provides systematic and sequential pressure changes to move fluid to intact lymphatic chains.
  Other Names: Flexi-touch Plus System
  Arms: Group I (pneumatic therapy, lymphedema management)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Voice Handicap Index-10 — Ancillary studies
  Other Names: VHI-10; Voice Handicap Index-10 (VHI-10)

SUMMARY:
This clinical trial tests whether adding the use of a pneumatic compression system with manual lymphatic drainage versus manual lymphatic drainage alone in treating patients with lymphedema after chemoradiation for stage II-IV head and neck cancer. Lymphedema can be the result of surgery, radiation therapy, chemotherapy or any combination of these procedures. Internal lymphedema has been shown to negatively affect speech production, swallowing, respiration, and voice. Flexitouch is an advanced pneumatic compression device (APCD) that consists of a 2-piece garment that provides pressure changes to move lymph fluid from the impaired area toward healthy regions of the body. Complete decongestive therapy (CDT) is standard of care for treating external lymphedema and involves manual lymphatic drainage (MLD) performed by licensed therapists followed by compression therapy. CDT has long been used for treating lymphedema of the limbs. Combining a pneumatic compression system with standard of care manual lymphatic drainage may have positive effects on speech, voice, and swallowing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare success rates in reducing internal and external lymphedema using manual lymphatic drainage (MLD) versus use of a pneumatic compression device (PCD). Assess efficacy of PCD and MLD.

II. Assess compliance of treatment in both groups. III. Assess changes in voice and swallowing in both groups.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I: Patients undergo 32 minute treatments twice daily for 12 weeks using the FlexiTouch Plus System and treatment with a lymphedema therapist weekly on weeks 2-11. Patients undergo nasolaryngoscopy and videofluoroscopic swallow study at baseline.

GROUP II: Patients undergo standard of care self-manual lymphatic drainage (technique instructions provided) twice daily for 12 weeks and treatment with a lymphedema therapist weekly on weeks 2-11. Patients undergo nasolaryngoscopy and videofluoroscopic swallow study at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Completed definitive chemoradiation for Stage II or greater, histologically proven cancer of the oral cavity, oropharynx, hypopharynx, pharynx or larynx with a curative intent
* Cognitive function adequate to understand and execute the elements of the protocol
* Willingness and ability to return to Mayo Clinic for follow-up care per protocol
* Resolution of acute dermatitis (skin must be intact without evidence of inflammation, infection or desquamation) as a result of chemoradiotherapy (CRT)
* Must demonstrate oropharyngeal competency that would allow some oral intake

Exclusion Criteria:

* Prior surgery, radiation, chemotherapy, or immunotherapy for head or neck cancer
* Acute radiation dermatitis, unhealed surgical wounds or surgical flap less than 2 months post-operative
* Acute facial infection
* Active congestive heart failure (CHF) or pulmonary edema
* Symptomatic carotid artery disease or bradycardia
* Increased intracranial pressure
* History of multiple cerebrovascular accidents (CVAs) or transient ischemic attacks (TIAs)
* > 50% internal carotid artery (ICA) blockage
* Upper quadrant deep vein thrombosis
* Known esophageal obstruction
* Percutaneous endoscopic gastrostomy (PEG) tube dependence with no oral intake
* Women of child-bearing potential
* (Active) pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-08-22 (Estimated); Study Completion 2024-08-22 (Estimated)

PRIMARY OUTCOMES:
Compare composite measurements of the face and neck for lymphatic drainage | Change from baseline and up to 12 weeks
  Will be completed at baseline and at the conclusion of the study to assess and compare the effects of traditional manual lymphatic drainage to those from use of a pneumatic compression system.
Change in lymphedema of the head and neck | Up to 12 weeks
  A reduction in one grade on the Mayo Clinic Lymphedema - head and neck (HN) Grading Scale (MCLGS) or one stage on the MD Anderson Cancer Center (MDACC) grading system for lymphedema of the head and neck.

SECONDARY OUTCOMES:
Improvements on quality of life (QOL) function | Up to 12 weeks
  Measured by QOL questionnaire and Facial and Neck Composite Measurements
  Status Scale:
  PSS-HN
Improvements on voice function | Up to 12 weeks
  Measured by Voice Handicap Index: VHI-10 and Consensus Aud- Perceptual Eval of Voice: CAPE-V
Improvements on swallowing function | Up to 12 weeks
  Measured by Videofluoroscopic Swallow Study, Functional Oral Intake Scale: FOIS, Eating Assessment Tool: EAT-10 and Performance

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Crujido, Principal Investigator — Mayo Clinic